CLINICAL TRIAL: NCT06958237
Title: Evaluation of Performance and Safety of the Medical Device: Salicylic Acid Wart Patch for the Treatment of Common Warts and Plantar Warts
Brief Title: Salicylic Acid Wart Patch for the Treatment of Common Warts and Plantar Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Langsteiner sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.1.
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Common Warts; Plantar Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients treated with wart patches (Experimental)
  Interventions: Device: salicylic acid wart patches

INTERVENTIONS:
Device: salicylic acid wart patches — The wart patches contain the auxiliary therapeutic substance salicylic acid at a concentration of 40%, which causes chemical exfoliation, removing the exfoliated skin. Salicylic acid softens the keratinised skin, making it easier to remove. The remedial process leads to the removal of the wart by exfoliation. The wart should disappear after about 7 days of using the patch. The treatment can be prolonged up to 21 days.
  The wart patch is intended for the treatment of common warts and plantar warts. The mechanism of action of the product is the barrier and protective action of the patch, reducing the possibility of spreading viral infection and, as an auxiliary, to exfoliate keratinised epidermis, accelerating the skin renewal process.

SUMMARY:
Common and plantar warts are a type of skin lesion caused by infection with the human papilloma virus. The incidence of warts is relatively high, with an estimated few to several per cent of the adult population affected. An even higher incidence of dermal warts is reported in the child and adolescent population, where it reaches nearly twenty per cent. The human papilloma virus (HPV) multiplies in the epidermal cells, leading to the formation of a skin lesion with a hyperkeratotic, uneven surface, called a wart. HPV infection can lead to various types of warts: including common warts, plantar warts, flat warts or condyloma acuminatum. Warts belong to skin lesions of a benign and self-limiting nature. Because of this, treatment of warts is often not applied. However, it is necessary to emphasise that warts, including in particular plantar warts, can be a source of pain as well as lead to psychological discomfort for the patient. Additionally, untreated warts are a potential source of subsequent infections.

For this reason, a variety of methods are used to treat warts, with the primary aim of removing the layer of diseased epidermis, as well as limiting the spread of the virus. The methods used to treat warts can be divided according to the nature of the agent used in the treatment - physical or chemical. Physical methods include cryotherapy, photodynamic therapy and surgical or laser wart removal. Chemical methods for the treatment of warts will be the use of ointments and solutions of substances such as salicylic acid, 5-fluorouracil, glycolic acid or purine acid. In addition, the treatment of warts also includes methods based on an occlusive action, involving the use of a barrier that shields the skin lesion and stops the spread of the virus.

This protocol concerns a study of salicylic acid wart patches. The aim of the study is to determine the efficacy and safety of their use in the treatment of common and plantar warts. The patches allow covering the lesion and the salicylic acid contained in them at a concentration of 40% has a keratolytic action allowing exfoliation of excessive epidermal proliferation caused by HPV infection. In addition, the mass of the product includes lanolin, which has an epidermal softening effect. The patches are intended for a patient population over six years of age, with common and plantar warts. The primary endpoints analysed in the study will be reduction in lesion size (assessed by dermatoscopic measurement), change in the number of warts in the area of the main wart-like lesion, occurrence of further dermal wart-like lesions in the treated area and incidence of adverse reactions. In addition, secondary endpoints to be analysed are reduction in lesion size (users' visual assessment), reduction in lesion visibility (users' visual assessment) and usability of the device.

ELIGIBILITY:
Inclusion Criteria:

* giving consent to participate in the clinical trial (consent of the minor's guardian where applicable);
* presence of at least 1 wart (common/plantar) on the body, with a lesion up to 1 cm in diameter;
* age, at least 6 years.

Exclusion Criteria:

* failure to meet at least 1 inclusion criterion;
* the patient has a known hypersensitivity to salicylic acid, salicylates or any other component of the patch;
* patients with renal impairment (renal failure);
* patients with skin conditions (e.g. inflammation, wounds, eczema) at the site of application,
* patients concurrently using other topical treatments in the area of the wart,
* diabetic patients.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
reduction in the size of the lesion | 30 minutes (single visit)
  reduction in the size of the lesion assessed by measuring with a dermatoscope
change in the number of warts in the area of the main wart-like lesion | 30 minutes (single visit)
  change in the number of warts in the area of the main wart-like lesion as assessed by the dermatologist
occurrence of further dermal wart-like lesions in the treated area | 30 minutes (single visit)
  occurrence of further dermal wart-like lesions in the treated area as assessed by the dermatologist
Adverse events | 30 minutes (single visit)
  Adverse events occuring during treatment of warts

SECONDARY OUTCOMES:
reduction in lesion size | 30 minutes (single visit)
  reduction in lesion size according to users' visual assessment
reduction in the visibility of the lesion | 30 minutes (single visit)
  reduction in the visibility of the lesion, user's visual assessment
usability of the device | 30 minutes (single visit)
  usability assessed with a questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Kowalska Clinic, Miechów, Lesser Poland Voivodeship, Poland